CLINICAL TRIAL: NCT06845748
Title: Assessment of Physical and Physiological Changes in Muscle Aging
Brief Title: Muscle Aging Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Matteo Bonato, Associate Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSR2023_BONATO
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Preventing Age-Related Muscle Loss: the Role of Exercise in Improving Strength, Function, and Well-being
Keywords: sarcopenia; aging; Frailty prevention; Exercise; interventional study
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity group (Experimental): Participants in this group will follow a structured physical activity program for 48 weeks. The intervention consists of muscle-strengthening sessions (bodyweight exercises at home) and aerobic sessions (moderate-intensity cardio exercise).
  The program is designed to improve muscle strength, mass, and function, aiming to counteract age-related muscle decline. Participants will undergo periodic assessments to measure physical performance, cognitive function, and quality of life.
  Interventions: Other: Physical activity Group
- Control Group (No Intervention): Participants in this group will not receive a structured exercise program. They will continue their usual lifestyle without specific physical activity recommendations.
  The control group will undergo the same periodic assessments as the experimental group to evaluate changes in muscle strength, function, body composition, and overall well-being over the 48-week study period.

INTERVENTIONS:
Other: Physical activity Group — This intervention consists of a 48-week structured physical activity program designed to counteract age-related muscle decline. Participants assigned to this group will engage in a home-based exercise program, including muscle-strengthening exercises (bodyweight exercises targeting major muscle groups; progressive difficulty based on individual capacity; designed for feasibility in daily life, requiring no specialized equipment) and aerobic exercise (moderate-intensity cardiovascular activity (e.g., brisk walking, cycling); target heart rate between 65-75% of the estimated maximum heart rate).
  The program follows guidelines from the American College of Sports Medicine (ACSM) and aims to improve muscle strength, function, and quality of life. It is distinct from other studies as it specifically targets preventing sarcopenia and muscle loss through a practical, home-based, and scalable intervention.
  Participants will be monitored through periodic assessments.
  Other Names: Exercise intervention
  Arms: Physical activity group

SUMMARY:
This study aims to assess the effects of physical activity in counteracting muscle aging. The increasing life expectancy worldwide has led to a rise in age-related muscle decline, which negatively impacts strength, function, and overall quality of life. Sedentary lifestyles further accelerate this process, increasing the risk of frailty, falls, fractures, and disability.

This randomized controlled trial (RCT) will investigate whether a structured exercise program can help reduce muscle deterioration. The study will involve 200 participants, divided into three age groups: i) Young adults (18-35 years); ii) Middle-aged adults (35-65 years); iii) Older adults (>65 years).

Participants will be assigned to either a physical activity intervention group or a control group. The intervention group will follow a 48-week structured program including, muscle-strengthening sessions (bodyweight exercises at home) and aerobic sessions (moderate-intensity cardio exercise). The control group will not receive any exercise prescription.

The primary objective is to evaluate whether physical activity improves muscle strength, measured through handgrip strength at 12 and 48 weeks.

Secondary objectives include: i) assessing changes in muscle mass, function, and quality of life; ii) measuring improvements in physical performance (aerobic capacity, balance, and mobility tests); iii) evaluating psychological and cognitive well-being.

This 48-week trial will consist of: i) baseline assessments (body composition, strength tests, physical and cognitive evaluations); ii) intervention period (12 weeks of structured training for the experimental group); iii) follow-up assessments (at 12 and 48 weeks).

All participants will undergo periodic evaluations, including anthropometric and body composition measurements (weight, BMI, muscle mass), aerobic and muscle strength tests (handgrip, knee extension, 1-rep max tests), functional mobility assessments (six-minute walking test, chair-stand test), psychological and cognitive evaluations (mood profiles, quality of life surveys, cognitive tests).

Engaging in regular exercise may help participants: i) maintain muscle mass and strength; ii) improve physical function and balance; iii) enhance overall well-being and independence; iv) reduce the risk of age-related disabilities.

Additionally, the study aims to provide valuable insights into the role of exercise in healthy aging, helping healthcare providers develop personalized interventions for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Must be able to engage in physical activity as prescribed in the study protocol.
* No pre-existing musculoskeletal conditions that would prevent safe participation.
* No history of hospitalization in the six weeks prior to enrollment.
* No acute or uncontrolled medical conditions that could interfere with exercise participation.
* Willing to sign an informed consent form before participation.

Exclusion Criteria:

* Severe Medical Conditions (cardiovascular diseases, severe respiratory diseases, neurological disorders)
* Cognitive and Psychological Conditions (severe cognitive impairment or dementia, psychiatric disorders)
* Pregnancy
* Use of anabolic or muscle-enhancing substances (use of steroids, testosterone therapy, or other performance-enhancing drugs within the past 6 months)
* Participation in ther Clinical Trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in handgrip strength at 12 and 48 weeks | Baseline, Week 12, and Week 48
  Handgrip strength will be measured using a hand dynamometer to assess the maximal isometric force of the dominant hand. The mean of three trials will be recorded, with 60-second rest intervals between attempts. An increase in handgrip strength over time will indicate the effectiveness of the physical activity intervention in maintaining or improving muscle function in aging adults.

SECONDARY OUTCOMES:
Change in muscle mass | Baseline, Week 12, and Week 48
  Body composition, including lean muscle mass, will be assessed using bioelectrical impedance analysis (BIA) to evaluate changes in muscle preservation and hypertrophy.
Change in Lower Limb Strength (Knee Extension Isometric Force, N) at 12 and 48 weeks | Baseline, Week 12, and Week 48
  Maximal isometric knee extension force will be measured using a dynamometer to assess improvements in lower limb muscle strength.
Change in Physical Performance (Six-Minute Walk Test, meters) at 12 and 48 weeks | Baseline, Week 12, and Week 48
  Walking endurance will be assessed using the Six-Minute Walk Test (6MWT) following the American Thoracic Society guidelines, measuring the total distance covered in six minutes.
Change in Functional Mobility (Chair Stand Test, repetitions) at 12 and 48 weeks | Baseline, Week 12, and Week 48
  The 30-second Chair Stand Test will evaluate lower limb strength and endurance by counting the number of times a participant can rise from a chair within 30 seconds.
Change in Balance and Postural Control (Mini-BESTest Score) at 12 and 48 weeks | Baseline, Week 12, and Week 48
  Balance and postural control will be measured using the Mini Balance Evaluation Systems Test (Mini-BESTest), which assesses postural adjustments, sensory orientation, and gait stability.
Change in Quality of Life (SF-12 Health Survey Score) at 12 and 48 weeks | Baseline, Week 12, and Week 48
  Quality of life will be assessed using the SF-12 questionnaire, which evaluates both physical and mental health components.
Change in Cognitive Function (Trail Making Test, A & B) at 12 and 48 weeks | Baseline, Week 12, and Week 48
  Executive function and processing speed will be evaluated using the Trail Making Test (TMT A & B), where participants connect numbered and lettered sequences as quickly as possible.
Change in Psychological Well-being (Profile of Mood States - POMS) at 12 and 48 weeks | Baseline, Week 12, and Week 48
  Mood states will be assessed using the Profile of Mood States (POMS) questionnaire, measuring anxiety, fatigue, vigor, depression, and confusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Milano, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jaeger J. Digit Symbol Substitution Test: The Case for Sensitivity Over Specificity in Neuropsychological Testing. J Clin Psychopharmacol. 2018 Oct;38(5):513-519. doi: 10.1097/JCP.0000000000000941. PMID 30124583
- [Background] Balsalobre-Fernandez C, Glaister M, Lockey RA. The validity and reliability of an iPhone app for measuring vertical jump performance. J Sports Sci. 2015;33(15):1574-9. doi: 10.1080/02640414.2014.996184. Epub 2015 Jan 2. PMID 25555023
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Seo DI, Kim E, Fahs CA, Rossow L, Young K, Ferguson SL, Thiebaud R, Sherk VD, Loenneke JP, Kim D, Lee MK, Choi KH, Bemben DA, Bemben MG, So WY. Reliability of the one-repetition maximum test based on muscle group and gender. J Sports Sci Med. 2012 Jun 1;11(2):221-5. eCollection 2012. PMID 24149193
- [Background] Lohman TG. Skinfolds and body density and their relation to body fatness: a review. Hum Biol. 1981 May;53(2):181-225. No abstract available. PMID 7239496
- [Background] Bisio A., Bove M. (2018) Cognitive Strategies to Enhance Motor Performance: Examples of Applying Action Observation, Motor Imagery and Psyching-up Techniques. Chapter 12 (pp. 248-281) of Handbook of Sport Neuroscience and Psychophysiology. Ed. Routledge.
- [Background] Sousa-Santos AR, Amaral TF. Differences in handgrip strength protocols to identify sarcopenia and frailty - a systematic review. BMC Geriatr. 2017 Oct 16;17(1):238. doi: 10.1186/s12877-017-0625-y. PMID 29037155